CLINICAL TRIAL: NCT06846762
Title: Real-world Study of DNA + RNA-NGS Co-testing in Patients with Driver Gene-negative, First-line Non-targeted Therapy-resistant Primary NSCLC (Dream Study)
Brief Title: DREAM Study: DNA/RNA-NGS Co-Testing in Driver-Negative, Treatment-Resistant NSCLC
Status: Recruiting | Type: Observational
Sponsor: Baohui Han (Other)
Responsible Party: Sponsor-Investigator, Baohui Han, director, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Other Study IDs: ShanghaiChestIS25009
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Primary Resistance; DNA+RNA-NGS; Driver Gene Testing; Targeted Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Formalin-Fixed Paraffin-Embedded (FFPE) samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Driver gene-positive patients with targeted therapy.: Patients who tested positive by DNA+RNA-NGS voluntarily choose to receive targeted therapy
  Interventions: Other: This study did not include intervention between the two cohorts
- Driver gene-positive patients without targeted therapy.: Patients who tested positive by DNA+RNA-NGS voluntarily choose to receive non-targeted therapy
  Interventions: Other: This study did not include intervention between the two cohorts

INTERVENTIONS:
Other: This study did not include intervention between the two cohorts — The study is divided into two parts, Part A and Part B. The purpose of Part A is to reveal the proportion of NSCLC patients who are primarily resistant to first-line non-targeted therapy due to the omission of driver genes (especially fusion variations) by DNA-NGS, the median PFS of patients in the first line, and clinical characteristics through synchronous co-testing of DNA and RNA NGS. The purpose of Part B is to compare the difference in ORR between patients with driver gene positivity identified through synchronous co-testing of DNA and RNA NGS who receive and do not receive targeted therapy, with subsequent treatment regimens determined at the discretion of the patients without any intervention measures.

SUMMARY:
The study is divided into two parts, Part A and Part B. The purpose of Part A is to reveal the proportion of NSCLC patients who are primarily resistant to first-line non-targeted therapy due to the omission of driver genes (especially fusion variations) by DNA-NGS, the median PFS of patients in the first line, and clinical characteristics through synchronous co-testing of DNA and RNA NGS. The purpose of Part B is to compare the difference in ORR between patients with driver gene positivity identified through synchronous co-testing of DNA and RNA NGS who receive and do not receive targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and above, male or female
2. Pathologically diagnosed with advanced or metastatic inoperable non-small cell lung cancer
3. Prior genetic testing [DNA-NGS] results show no mutations in EGFR, BRAF, MET, HER2, KRAS, FGFR2/3，no amplifications in MET and HER2 and no fusions in ALK, ROS1, RET, NTRK, NRG1, EGFR, MET, BRAF, FGFR2/3
4. Based on negative driver gene results, received first-line non-targeted therapy with rapid progression or intolerance, with a progression-free survival (PFS) of ≤6 months (regardless of drug exposure time, calculated from the first day of medication)
5. Have retained tumor tissue samples prior to first-line treatment
6. Patients are from medical centers that can ethically affiliate and have accessible clinical follow-up data.

Exclusion Criteria:

1. Patients who do not meet any of the necessary inclusion criteria
2. Presence of other pulmonary diseases that require treatment or are severe, including but not limited to active pulmonary tuberculosis, interstitial lung disease, etc.
3. Presence of active infections that require systemic treatment
4. History of drug abuse or alcohol abuse, or mental illness, or suspected allergy or intolerance to the study drug or any of its components
5. Any other conditions deemed unsuitable for entry into this study by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NSCLC patients who are primarily resistant to first-line non-targeted therapy due to the omission of driver genes (especially fusion variations) by DNA-NGS.
Sampling Method: Non-Probability Sample
Enrollment: 508 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with advanced or metastatic inoperable NSCLC who test positive for driver genes upon re-testing with DNA+RNA NGS | 2026.1
ORR | 2027.1

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes